CLINICAL TRIAL: NCT01671995
Title: Optimising Congestive Heart Failure Outpatient Clinic Project (OPTIMAL)
Brief Title: Optimising Congestive Heart Failure Outpatient Clinic Project
Acronym: OPTIMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Thomas Kahan, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIMAL
Record Dates: First submitted 2012-08-19; First posted 2012-08-24 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Heart Failure
Keywords: Heart failure; Quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse monitored heart failure program (Experimental): To assess whether a nurse monitored management programme at the hospital outpatient clinic would improve quality of life, as compared to standard primary health care.
  Interventions: Procedure: Nurse monitored heart failure program
- Standard primary health care (Active Comparator): To assess whether a nurse monitored management programme at the hospital outpatient clinic would improve quality of life, as compared to standard primary health care.
  Interventions: Procedure: Standard primary health care

INTERVENTIONS:
Procedure: Nurse monitored heart failure program — Standard program for a heart failure clinic with information, education, drug titration
  Arms: Nurse monitored heart failure program
Procedure: Standard primary health care — Standard care in primary care according to national guidelines but at the discretion of the primary care caregiver
  Arms: Standard primary health care

SUMMARY:
This study examines whether a nurse monitored management program at the hospital heart failure outpatient clinic can improve quality of life in elderly patients with chronic heart failure, as compared to standard treatment in primary healthcare.

DETAILED DESCRIPTION:
Patients 60 years of age or more hospitalized with heart failure according to New York Heart Association (NYHA) class II-IV and systolic dysfunction (left ventricular ejection fraction less than 0.45) are investigated before discharge and than randomized to the nurse monitored management program or to standard care. Examinations are performed at 0, 6, 12, and 18 months, and include clinical signs and symptoms, quality of life, biochemical assessment, echocardiography and drugs used. The study will be completed when all patients have passed the 18 month follow up examination. Quality of life is assessed by the Nottingham health profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years of age or older
* Hospitalized with heart failure according to New York Heart Association (NYHA) class II-IV
* Left ventricular systolic dysfunction with an ejection fraction below 0.45, by echocardiography

Exclusion Criteria:

* An acute myocardial infarction or unstable angina pectoris within the last three months
* Valvular stenosis
* Dementia
* Severe concomitant disease
* Refusal to participate.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 1996-01; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Quality of life | 18 months
  Nottingham health profile used for quality of life assessment

SECONDARY OUTCOMES:
Hospitalizations | 18 months
  Registry data that cover all hospitalizations for all patients
Evaluation of heart failure medication | 18 months
  Whether patients receive appropriate drug therapy (drug classes) and reach target doses of heart failure medication
Mortality | 18 months
  Mortality from death certificates obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Edner, MD, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Danderyd University Hospital Corp, Stockholm, Sweden

REFERENCES:
- [Result] Mejhert M, Kahan T, Persson H, Edner M. Limited long term effects of a management programme for heart failure. Heart. 2004 Sep;90(9):1010-5. doi: 10.1136/hrt.2003.014407. PMID 15310688
- [Result] Mejhert M, Linder-Klingsell E, Edner M, Kahan T, Persson H. Ventilatory variables are strong prognostic markers in elderly patients with heart failure. Heart. 2002 Sep;88(3):239-43. doi: 10.1136/heart.88.3.239. PMID 12181213
- [Result] Mejhert M, Kahan T, Persson H, Edner M. Predicting readmissions and cardiovascular events in heart failure patients. Int J Cardiol. 2006 Apr 28;109(1):108-13. doi: 10.1016/j.ijcard.2005.07.015. Epub 2005 Oct 5. PMID 16213040
- [Result] Mejhert M, Kahan T, Edner M, Persson HE. Sex differences in systolic heart failure in the elderly: the prognostic importance of left ventricular mass in women. J Womens Health (Larchmt). 2008 Apr;17(3):373-81. doi: 10.1089/jwh.2007.0487. PMID 18338962